CLINICAL TRIAL: NCT06770517
Title: Defeating Fear With Exposure Therapy Delivered by Mental Health Nurses in Primary Care for Anxiety Disorders in Older Adults - a Cluster-randomised Controlled Trial
Brief Title: Exposure Therapy for Late-life Anxiety
Acronym: DeFEAD65+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProPersona (Other)
Collaborators: Radboud University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Gert-Jan Hendriks, prof.dr., ProPersona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL87105.091.24; 10390022210020 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-12-11; First posted 2025-01-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Anxiety Disorders; Anxiety Depression
Keywords: exposure therapy; anxiety disorders; older adults; late-life anxiety; primary care
MeSH Terms: conditions — Anxiety Disorders | interventions — Implosive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: First assessments will be applied by project researchers and the following assessments will be applied by independent research assistants who are blinded for the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exposure therapy (Experimental): The participants will receive exposure therapy, entailing 8 sessions of 30 minutes spread over 12 weeks. The first session is 60 minutes long. The exposure therapy will be match to the needs and symptoms of the participant.
  Interventions: Behavioral: Exposure therapy
- Usual Care group (Active Comparator): This group will receive the usual care given by GP's based on the Nederlands Huisartsen Genootschap (NHG) standard practice in the Netherlands for anxiety disorders.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Exposure therapy — The exposure therapy will be given by the mental health care nurses (MHN) working in primary care centres. In addition, there will be eight sessions spread over 12 weeks. The first session will be 60 minutes long and the rest will be 30 minutes long.
  Other Names: Cognitive behavioral therapy
  Arms: Exposure therapy
Behavioral: Usual Care — The Usual Care group will receive care based on the general practitioners guidelines for anxiety disorders in the primary care center. This will entail possible medication, e-learning or psycho-education, problem solving therapy or a referral to a mental health institution.
  Arms: Usual Care group

SUMMARY:
The primary objective is to evaluate the (cost-)effectiveness of exposure therapy (ET) delivered by trained mental health nurses (MHNs) in terms of anxiety symptoms and quality of life for late life anxiety disorders in primary care compared to usual care (UC).

UC is not restricted, and the general practitioner (GP) is encouraged to work according to the guidelines of the Dutch College of GPs.

Participants in the ET group will receive 30-minute ET sessions delivered by a trained mental health nurse, during 8 sessions within the span of 12 weeks. Participants will fill in questionnaires before, during and after treatment, with a 1-year follow-up. The main study parameters are anxiety severity, quality of life and societal costs.

DETAILED DESCRIPTION:
Rationale: Anxiety disorders are common and have a high disease burden throughout the life span. Nonetheless, older people with anxiety disorders remain undiagnosed and thus undertreated. Ageism, changes in symptom phenomenology at older age and transportation barriers are reasons for underdiagnosis/-treatment. Moreover, when treated, older patients generally receive pharmacotherapy, while adverse effects increase with age and 75% of older persons prefer psychotherapy. The most effective psychotherapy, i.e. exposure therapy, has not yet been evaluated for older adults with anxiety in primary care.

Exposure Therapy (ET) is the most effective intervention for all anxiety disorders in adults. It has the potential to reduce the risk of chronicity, inappropriate healthcare use, inappropriate drug use, and unnecessary referral to specialist mental healthcare providers, which often include long, costly treatment trajectories. Exposure is well-suited to be delivered by mental health nurses (MHNs; or POH-GGZ (praktijkondersteuner geestelijke gezondheidszorg) in Dutch) in primary care centers (PCCs) because older people visit their general practitioner (GP) regularly, and PCCs in the Netherlands have the availability of MHNs. However, they are currently not equipped to offer exposure. Introducing MHN-led exposure is likely to be (cost-)effective as it matches patients' preferences and prevents inadequate or costly treatments.

Objective: The primary objective is to evaluate the (cost-)effectiveness of ET delivered by trained MHNs regarding anxiety symptoms and quality of life for late-life anxiety disorders in primary care compared to Usual Care (UC). UC is not restricted, and the GP is encouraged to work according to the guidelines of the Dutch College of GPs.

Study design: A multi-center cluster-randomized controlled trial (RCT) with two parallel groups: a) ET and b) UC, in PCCs with a 1-year follow-up.

Study population: 170 patients, 65 years and older, with an anxiety disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

Intervention (if applicable): During 8 sessions within the span of 12 weeks, 30-minute ET sessions are delivered by a trained mental health nurse.

Main study parameters/endpoints: Anxiety severity as assessed with the Geriatric Anxiety Inventory (GAI), societal costs with the Trimbos and iMTA(Institute for Medical Technology Assessment) questionnaire on Costs associated with Psychiatric illness (TIC-P) and quality of life using the EuroQol 5 Dimension 5 Level version (EQ-5D-5L) during the 12-week treatment period and 1-year follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Though the burden includes investment of the patient, no risks are associated with participation in the study. By offering participants ET in the PCC by the MHN, the participants will benefit immediately as we expect a positive influence on their anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 anxiety disorder using the Mini Internationaal Neuropsychiatrisch Interview (MINI).
* One of the following DSM-5 anxiety disorders will be diagnosed, Generalized Anxiety Disorder, Agoraphobia, Panic Disorder or Social Anxiety Disorder.
* Participants are required to be sufficient in Dutch.

Exclusion Criteria:

* Exclusion criteria include somatic and/or another psychiatric morbidity that could interfere with diagnosing or treatment.
* Moderate to severe suicidality, which will be determined using the MINI
* Chronic and interfering substance or alcohol abuse
* Having received previous psychotherapy including exposure in the past year. -
* Antidepressants and benzodiazepines use are allowed if on a stable dose for a minimum of 8 weeks.
* Participants will be excluded if they score lower than 18 points on the MoCa (115). A score of <18 is indicative for moderate to severe cognitive impairment. - Participants will be excluded if they are terminally ill.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-06-23 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Is ET performed by MHNs effective compared to UC in primary care for older adults with anxiety disorders in terms of QUALYs and symptoms of anxiety? | Pre-intervention, post-intervention (after 12 weeks of treatment), 3-month follow-up (FU), 6- month FU, 9-month FU, 12-month FU
  1. Anxiety severity will be assessed with the Geriatric Anxiety Inventory (GAI). The GAI is a self-report measure of general anxiety symptoms over the last week. Total scores range from 0-20, with higher scores indicating greater anxiety.
  2. The second questionnaire used is the EuroQol 5-Dimension 5-Level version (EQ-5D-5L), which is used to measure quality of life. It has five subscales consisting of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 3L classification system defines the 243 health states by combining different levels (one from each dimension), ranging from 11111 (full health) to 33333 (worst health). The 5L classification system comprises the same five dimensions as the 3L, but each dimension has two more levels to the existing three levels. Accordingly, the 5L system defines the 3,125 health states ranging from 11111 to 55555.
  Both questionnaires will be used during the 12-week treatment period and during the 1-year follow-up.
Is ET performed by MHNs cost-effective compared to UC in primary care for older adults with anxiety disorders in terms of QUALYs and symptoms of anxiety? | Pre-intervention T0, post-intervention (after 12 weeks of treatment, also knows as T9), 3-month FU, 6- month FU, 9-month FU, 12-month FU
  The aim is to relate the incremental costs of ET compared with UC to the incremental health effects. Both a cost-effectiveness analysis (CEA) and a cost-utility analysis (CUA) will be performed from a societal and healthcare perspective.
  1. For the cost-effectiveness analysis Quality-Adjusted Life-Years (QUALYs) will be assessed with the EQ-5D-5L.
  2. Anxiety severity will be assessed with the Geriatric Anxiety Inventory (GAI). Total scores range from 0 to 20, with higher scores indicating greater anxiety.
  3. To assess societal costs, the TIC-P will be used. This questionnaire is the modified version of the Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TiC-P). Cost categories that will be included are: 1) healthcare costs; 2) lost productivity costs; 3) patient costs. Valuation will be done according to Dutch costing guidelines. Higher scores indicate higher societal costs.

SECONDARY OUTCOMES:
Are there differences regarding secondary outcomes, such as disorder specific anxiety symptoms, comorbid depressive symptoms, general functioning and the use of psychoactive medications (i.e., antidepressants and benzodiazepines) between ET and UC? | Pre-intervention T0, post-intervention (12-week), 3-month FU, 6- month FU, 9-month FU, 12-month FU
  1. Social Anxiety: Liebowitz Social Anxiety Scale (LSAS), total score ranging 0-144.
  2. Generalized Anxiety Disorder (GAD): GAD-7 scale, total score ranging 0-21. 3) Panic Disorder: Panic Disorder Severity Scale-Self Report (PDSS-SR), total score ranging 0-28.
  For all three questionnaires is a higher score an indication for more severe anxiety.
  4) Agoraphobia: Mobility Inventory (MI), 27 items rated from 0 (never avoids) to 4 (always avoids). Scores are averaged based on situations experienced alone or accompanied.
  Depressive Symptoms: Quick Inventory of Depressive Symptoms (QIDS-SR), total score ranging 0-27. Higher scores indicate greater severity.
  General Functioning: 12-item World Health Organization Disability Assessment Schedule (WHODAS 2.0). Average scores 1 (no disability) to 5 (extreme disability).
  Medication use: use of benzodiazepines and antidepressants, binary yes/no.

OTHER OUTCOMES:
Do factors such as ageist biases of participants and mental health nurses, cognitive functioning, therapeutic expectations and alliance influence the effectiveness of exposure therapy in treating late-life anxiety? | Pre-intervention T0, post intervention (after 12 weeks of treatment, also knows as T9) and at the 12 month follow-up
  * Ageist biases of participants and mental health nurses will be measured using the 12-item Shortened Expectations Regarding Aging Survey (ERA-12), consisting of 3 subscales and total score ranging 0 to 100.
  * Cognitive functioning will be measured with Montréal Cognitive Assessment scale (MoCA) total score ranging 0-30.
  * Therapeutic expectations will be measured with Credibility & Expectancy Questionnaire with 6 items. This measure is scored on a Likert scale ranging from 1 to 9 (e.g., 1 means 'not at all', 5 'somewhat', and 9 'very much') or from 0% to 100% (in 10-point increments). Items 4 and 6, coded from 0%-100%, are converted linearly on a Likert scale from 1 to 9.
  * Therapeutic alliance will be measured with Working Alliance Inventory (WAI), total score is the average of 12 items, with a maximum score of 5.
Do changes in threat expectancy, avoidance and safety behaviours, self-efficacy, metacognitions (i.e. beliefs about cognition) and worry partially explain the effectiveness of ET compared to UC | Pre-intervention T0, during intervention, post intervention (after 12 weeks of treatment, also knows as T9) and at the 12 month follow-up
  - Threat expectancy: As part of the treatment protocol, participants rate: Before exposure: Threat expectancy (0-100%) - likelihood of feared outcome. After exposure: Threat occurrence (0-100%) - extent of feared outcome, and Adjusted threat expectancy (0-100%) - likelihood of outcome if repeated.
  * Avoidance will be measured with:
    1. Brief Experiential Avoidance Questionnaire (BEAQ), 15 items, rated 1-6.
    2. The Cognitive-Behavioural Avoidance Scale (CBAS), 31 items, rated 1-5, measuring different types of avoidance.
  * Safety Behaviours: Safety Behaviour Scale (SBS), 14 items, rated 0-4.
  * Self-Efficacy: General Self-Efficacy Scale (GSE), total score 10-40. Higher scores indicate greater self-efficacy.
  Metacognitions: Metacognition Questionnaire-30 (MCQ-30), total score 30-120. Higher scores indicate more unhelpful metacognitions.
  Worry: Assessed with the Penn State Worry Questionnaire (PSWQ), 16 items, rated 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique NJ Rijkelijkhuizen, MSc, Study Chair — ProPersona; Özge Baturlar, MSc, Study Chair — ProPersona
Locations (1):
- RadboudUMC, Nederland, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sullivan SD, Mauskopf JA, Augustovski F, Jaime Caro J, Lee KM, Minchin M, Orlewska E, Penna P, Rodriguez Barrios JM, Shau WY. Budget impact analysis-principles of good practice: report of the ISPOR 2012 Budget Impact Analysis Good Practice II Task Force. Value Health. 2014 Jan-Feb;17(1):5-14. doi: 10.1016/j.jval.2013.08.2291. Epub 2013 Dec 13. PMID 24438712
- [Background] Craske MG, Treanor M, Zbozinek TD, Vervliet B. Optimizing exposure therapy with an inhibitory retrieval approach and the OptEx Nexus. Behav Res Ther. 2022 May;152:104069. doi: 10.1016/j.brat.2022.104069. Epub 2022 Mar 15. PMID 35325683
- [Background] Knowles KA, Tolin DF. Mechanisms of Action in Exposure Therapy. Curr Psychiatry Rep. 2022 Dec;24(12):861-869. doi: 10.1007/s11920-022-01391-8. Epub 2022 Nov 18. PMID 36399234
- [Background] Yochim BP, Mueller AE, Segal DL. Late life anxiety is associated with decreased memory and executive functioning in community dwelling older adults. J Anxiety Disord. 2013 Aug;27(6):567-75. doi: 10.1016/j.janxdis.2012.10.010. Epub 2012 Nov 6. PMID 23298889
- [Background] Buchholz JL, Abramowitz JS. The therapeutic alliance in exposure therapy for anxiety-related disorders: A critical review. J Anxiety Disord. 2020 Mar;70:102194. doi: 10.1016/j.janxdis.2020.102194. Epub 2020 Jan 18. PMID 32007734
- [Background] Saif-Ur-Rahman KM, Mamun R, Eriksson E, He Y, Hirakawa Y. Discrimination against the elderly in health-care services: a systematic review. Psychogeriatrics. 2021 May;21(3):418-429. doi: 10.1111/psyg.12670. Epub 2021 Feb 26. PMID 33634922
- [Background] Wuthrich VM, Meuldijk D, Jagiello T, Robles AG, Jones MP, Cuijpers P. Efficacy and effectiveness of psychological interventions on co-occurring mood and anxiety disorders in older adults: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2021 Jun;36(6):858-872. doi: 10.1002/gps.5486. Epub 2021 Jan 2. PMID 33368598
- [Background] Hendriks GJ, Kampman M, Keijsers GP, Hoogduin CA, Voshaar RC. Cognitive-behavioral therapy for panic disorder with agoraphobia in older people: a comparison with younger patients. Depress Anxiety. 2014 Aug;31(8):669-77. doi: 10.1002/da.22274. Epub 2014 May 27. PMID 24867666
- [Background] Jayasinghe N, Finkelstein-Fox L, Sar-Graycar L, Ojie MJ, Bruce ML, Difede J. Systematic Review of the Clinical Application of Exposure Techniques to Community-Dwelling Older Adults with Anxiety. Clin Gerontol. 2017 May-Jun;40(3):141-158. doi: 10.1080/07317115.2017.1291546. Epub 2017 Feb 6. PMID 28452667
- [Background] Abramowitz JS. The practice of exposure therapy: relevance of cognitive-behavioral theory and extinction theory. Behav Ther. 2013 Dec;44(4):548-58. doi: 10.1016/j.beth.2013.03.003. Epub 2013 Mar 13. PMID 24094780
- [Background] Beesdo-Baum K, Jenjahn E, Hofler M, Lueken U, Becker ES, Hoyer J. Avoidance, safety behavior, and reassurance seeking in generalized anxiety disorder. Depress Anxiety. 2012 Nov;29(11):948-57. doi: 10.1002/da.21955. Epub 2012 May 11. PMID 22581482
- [Background] Benitez CI, Smith K, Vasile RG, Rende R, Edelen MO, Keller MB. Use of benzodiazepines and selective serotonin reuptake inhibitors in middle-aged and older adults with anxiety disorders: a longitudinal and prospective study. Am J Geriatr Psychiatry. 2008 Jan;16(1):5-13. doi: 10.1097/JGP.0b013e31815aff5c. PMID 18165458
- [Background] Schuurmans J, Comijs HC, Beekman AT, de Beurs E, Deeg DJ, Emmelkamp PM, van Dyck R. The outcome of anxiety disorders in older people at 6-year follow-up: results from the Longitudinal Aging Study Amsterdam. Acta Psychiatr Scand. 2005 Jun;111(6):420-8. doi: 10.1111/j.1600-0447.2005.00531.x. PMID 15877708
- [Background] Mohlman J. A community based survey of older adults' preferences for treatment of anxiety. Psychol Aging. 2012 Dec;27(4):1182-90. doi: 10.1037/a0023126. Epub 2011 Apr 4. PMID 21463061
- [Background] Kessler EM, Blachetta C. Age cues in patients' descriptions influence treatment attitudes. Aging Ment Health. 2020 Jan;24(1):193-196. doi: 10.1080/13607863.2018.1515889. Epub 2018 Oct 31. PMID 30380336
- [Background] Wolitzky-Taylor KB, Castriotta N, Lenze EJ, Stanley MA, Craske MG. Anxiety disorders in older adults: a comprehensive review. Depress Anxiety. 2010 Feb;27(2):190-211. doi: 10.1002/da.20653. PMID 20099273
- [Background] van Balkom AJ, Beekman AT, de Beurs E, Deeg DJ, van Dyck R, van Tilburg W. Comorbidity of the anxiety disorders in a community-based older population in The Netherlands. Acta Psychiatr Scand. 2000 Jan;101(1):37-45. doi: 10.1034/j.1600-0447.2000.101001037.x. PMID 10674949
- [Background] Hohls JK, Konig HH, Raynik YI, Hajek A. A systematic review of the association of anxiety with health care utilization and costs in people aged 65 years and older. J Affect Disord. 2018 May;232:163-176. doi: 10.1016/j.jad.2018.02.011. Epub 2018 Feb 15. PMID 29494900
- [Background] Hendriks GJ, Janssen N, Robertson L, van Balkom AJ, van Zelst WH, Wolfe S, Oude Voshaar RC, Uphoff E. Cognitive behavioural therapy and third-wave approaches for anxiety and related disorders in older people. Cochrane Database Syst Rev. 2024 Jul 8;7(7):CD007674. doi: 10.1002/14651858.CD007674.pub3. PMID 38973756
- [Background] Janssen NP, Lucassen P, Huibers MJH, Ekers D, Broekman T, Bosmans JE, Van Marwijk H, Spijker J, Oude Voshaar R, Hendriks GJ. Behavioural Activation versus Treatment as Usual for Depressed Older Adults in Primary Care: A Pragmatic Cluster-Randomised Controlled Trial. Psychother Psychosom. 2023;92(4):255-266. doi: 10.1159/000531201. Epub 2023 Jun 29. PMID 37385226
- See also: DeFEAD65+ is based on the BEATDeP (Behavioural activation for depression among older adults) study — https://link.springer.com/article/10.1186/s12888-017-1388-x